CLINICAL TRIAL: NCT01737021
Title: A Psycho-educational Intervention to Improve Family Mental Health and Child Educational Outcomes Following Admission to PICU: A Pilot Study
Brief Title: Improving Outcomes After PICU Admission: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Children of St Mary's Intensive Care (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CRO2015
Record Dates: First submitted 2012-11-01; First posted 2012-11-29 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Critical Illness
Keywords: PICU; Critical illness; Outcomes; Mental health; Education; Randomized Controlled Trial (RCT); Pilot; Feasibility
MeSH Terms: conditions — Critical Illness; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psycho-educational intervention (Experimental): Psycho-education
  Interventions: Other: Psycho-education
- Treatment as usual (No Intervention)

INTERVENTIONS:
Other: Psycho-education — The information given to parents will cover expected reactions that follow a PICU admission; how parents can help their child cope with these reactions; how to recognise warning signs; and sign-posting of appropriate follow-up services (if relevant). There will also be a follow-up telephone call to reinforce the information and to support parents in putting it in to practice, if appropriate.
  Arms: Psycho-educational intervention

SUMMARY:
1. Evaluate the feasibility and acceptability of an information based intervention delivered to parents following their child's admission to paediatric intensive care;
2. Evaluate the feasibility and acceptability of the study design and procedures;
3. Explore the effects of the intervention on parent and child psychological outcomes 3-6 months post discharge from PICU;
4. Explore the effects of parental stress experienced during PICU admission on the effectiveness of the intervention;
5. To provide data that, combined with results from other studies, could inform the sample size for a future multi-site RCT.

DETAILED DESCRIPTION:
Most children are now expected to make a complete medical recovery following admission to PICU. However, research suggests that some children will go on to develop psychological difficulties, such as problems with emotions, behaviour, and learning. In addition, parents themselves may suffer with emotional difficulties. Although the follow-up of survivors is recommended, there are currently no specific guidelines in place. Intervention in the early stages of recovery could help families pull through without long lasting after-effects.

ELIGIBILITY:
Inclusion Criteria:

* Unplanned emergency admissions to PICU for at least 12 hours
* Parent or primary carer speaks and can read English

Exclusion Criteria:

* Child dies whilst on ward
* Child discharged with a terminal illness
* Child has had multiple PICU admission in the past
* Staff feel it is inappropriate to approach family
* Family live overseas

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2012-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Garralda, M.D., Principal Investigator — Imperial College London

REFERENCES:
- [Derived] Als LC, Nadel S, Cooper M, Vickers B, Garralda ME. A supported psychoeducational intervention to improve family mental health following discharge from paediatric intensive care: feasibility and pilot randomised controlled trial. BMJ Open. 2015 Dec 29;5(12):e009581. doi: 10.1136/bmjopen-2015-009581. PMID 26715482

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment as Usual: There is no existing standard follow up for parents of children discharged from PICU.
Period: Overall Study
Arm/Group | Psycho-educational Intervention | Treatment as Usual
Started | 22 | 9
Completed | 17 | 6
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Psycho-educational Intervention: Received psycho-educational intervention.
- Total: Total of all reporting groups
Arm/Group | Psycho-educational Intervention | Treatment as Usual | Total
Number analyzed (Participants) | 17 | 6 | 23
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 6.00 [5.50 to 10.50] | 9.00 [5.50 to 11.00] | 6.00 [6.00 to 11.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: The Number of Feasibility Criteria Successfully Met
Description: Feasibility success criteria have been defined a priori for the intervention and study design. There are six feasibility criteria related to the intervention, covering aspects of the timing of the intervention, compliance, and evaluation. There are also six feasibility criteria related to the study design, covering recruitment rate; participation rate; acceptability of procedures; attrition rate; and the time-scale of data collection.
  Dependent on the number of criteria successfully met, the following classification will be used:
  "*" 0-2/6 criteria met - Stop; intervention and/or study design not feasible. "*" 3-4/6 criteria met - Continue with modifications; feasible intervention and/or study design with modifications.
  "*" 5/6 criteria met - Continue without modifications, but monitor closely; feasible intervention and/or study design with close monitoring.
  "*" 6/6 criteria met - Continue without modifications; feasible intervention and/or study design as is.
Time Frame: 3-6 months post discharge from PICU
Measure: Number; unit: Number of criteria successfully met
Groups:
- Intervention: There were six feasibility criteria related to the intervention, covering aspects of the timing of the intervention, compliance, and evaluation.
- Study Design: There were also six feasibility criteria related to the study design, covering recruitment/ participation rate, acceptability of procedures, loss to follow-up rate, and the time-scale of data collection.
Arm/Group | Intervention | Study Design
Number analyzed (Participants) | 17 | 23
Number of criteria successfully met | 3 | 1

2. Secondary Outcome: Impact of Events Scale (IES)
Description: Validated measure of post-traumatic stress symptoms in the parent.
Time Frame: 3-6 months post discharge from PICU
Reporting Status: Not Posted

3. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS)
Description: Validated measure of anxiety and depression in the parent.
Time Frame: 3-6 months post discharge from PICU
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Psycho-educational Intervention | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/9
Other Adverse Events (participants affected / at risk) | 0/22 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes